CLINICAL TRIAL: NCT06975046
Title: Aerodynamic Measurements in the Pediatric Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: University of Iowa (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024-1776; A539770 (Other: UW Madison); SMPH/SURGERY/OTOLARYNGOLOGY (Other: UW Madison); Protocol Version 11/20/2024 (Other: UW Madison); 1R01DC021415 (NIH)
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-05

CONDITIONS: Normal Voice

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Complete airflow interruption (Experimental)
  Interventions: Device: Complete airflow interruption
- Incomplete airflow interruption (Experimental)
  Interventions: Device: Incomplete airflow interruption
- Airflow redirection (Experimental)
  Interventions: Device: Airflow redirection

INTERVENTIONS:
Device: Complete airflow interruption — Participants will produce a sustained vowel into a mouthpiece (with nose-clip) connected to a PVC tube, with a balloon valve
  Arms: Complete airflow interruption
Device: Incomplete airflow interruption — Incomplete airflow interruption uses a Y-shaped device. The participant produces a sustained /a/ into a mouthpiece and air filter connected to the tube. The tube splits into two tubes distally.
  Arms: Incomplete airflow interruption
Device: Airflow redirection — Participant phonates through a mouthpiece into a PVC tube that splits into two paths. One path is connected to an open balloon valve. When the balloon is inflated and blocks the path, air is redirected into the other path which is gated by a one-way valve.
  Arms: Airflow redirection

SUMMARY:
The goal of this clinical trial is to create a vocal health database of people aged 4-17 with no diagnosed voice pathology. The main question it aims to answer is:

* what is the best way to assess pediatric voices; and,
* what are the differences between healthy and dysphonic pediatric voices?

Participants will complete one 60 minute session involving one of three types of aerodynamic interruption.

DETAILED DESCRIPTION:
The primary goals of this research are to develop noninvasive aerodynamic assessments specific to the pediatric population, and to describe differences between healthy and dysphonic pediatric voices between the ages of 4-17 years. To account for challenges associated with pediatric data collection, we will modify our current devices and methods of aerodynamic assessment to be better suited for use with the pediatric population and aim to increase measurement reliability in younger subjects. Our proposed modifications include shorter trial times, auditory masking, the use of cheek restraints, and gamification.

After identification of optimal data collection conditions for each method, we will compare these in a large group of children with normal voice. These data will be compared to data from children with vocal fold nodules or polyp. All data will be compiled into a pediatric vocal health database

ELIGIBILITY:
Inclusion Criteria - Healthy Control:

* Age 4-17 years
* Normal voice
* No history of voice or other pertinent health disorders

Exclusion Criteria - Healthy Control:

* Neuromuscular disorder affecting the larynx
* History of respiratory or laryngeal disease
* History of smoking
* Hearing impairment
* Cognitive impairment that might impact ability to perform the tasks required by the study

Inclusion Criteria - Abnormal Voice:

* Age 4-17
* Laryngeal pathology

Exclusion Criteria - Abnormal Voice:

* No laryngeal disorder

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 365 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Compare subglottic pressure across different airflow interruption methods | 60 minutes
  Subglottic pressure is measured in kPa of leakage of air between the vocal folds and the resistance to that flow during speech
Compare phonation threshold pressure (PTP) across airflow interruption methods | 60 minutes
  PTP is is calculated by subtracting the intraoral pressure at phonation cessation from the subglottal pressure (Ps).
Compare laryngeal resistance across airflow interruption methods | 90 minutes
  Pressure and airflow measurements can be taken and entered into equations (Ps = (LR) U1+ Z1U1 and Ps = (LR)U2+Z2U2) to calculate Laryngeal resistance and Ps.
Compare subglottic pressure between benign vocal fold lesions and normal voices | 90 minutes
  Subglottic pressure is measured in kPa of leakage of air between the vocal folds and the resistance to that flow during speech
Compare PTP between benign vocal fold lesions and normal voices | 90 minutes
  PTP is is calculated by subtracting the intraoral pressure at phonation cessation from the subglottal pressure (Ps).
Compare laryngeal resistance between benign vocal fold lesions and normal voices | 90 minutes
  Pressure and airflow measurements can be taken and entered into equations (Ps = (LR) U1+ Z1U1 and Ps = (LR)U2+Z2U2) to calculate Laryngeal resistance and Ps.
Compare vocal efficiency between benign vocal fold lesions and normal voices | 90 minutes
  Vocal efficiency is calculated using aerodynamic to acoustic power.
Compare mean airflow rate between benign vocal fold lesions and normal voices | 90 minutes
  Mean airflow (I) = Ps / laryngeal resistance (Lr).

CONTACTS AND LOCATIONS:
Overall Officials: Jack Jiang, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - University of Wisconsin - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes